CLINICAL TRIAL: NCT05774821
Title: Surgical Treatment of Tricuspid Valve Regurgitation in Patients With Cardiac Implantable Electronic Devices: Long Term Results
Status: Completed | Type: Observational
Sponsor: Michele De Bonis (Other)
Responsible Party: Sponsor-Investigator, Michele De Bonis, Chief of Cardiac Surgery of Advanced and Research Therapies, Ospedale San Raffaele
Organization: Ospedale San Raffaele (Other)
Other Study IDs: TR-CIED-LTR
Record Dates: First submitted 2023-01-30; First posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Tricuspid valve surgery — Surgical repair or valve prosthesis implant to treath the regurgitation of the tricuspid valve

SUMMARY:
Old trials aimed to evaluate Implantable Cardioverter-Defibrillator (ICD) safety and efficacy demonstrated a meaningful decreased rates of sudden death but an increased rate of hospitalization for heart failure . At the time, the chance that an endocardial lead could cause a significant tricuspid regurgitation (TR), leading to worsening heart failure, was not widely considered. Whereas, it is now well established that in patients with cardiac implantable electronic device (CIEDs), moderate or severe TR occurs frequently and it is associated with increased mortality and hospitalization for heart failure.

The present study aims to report the long-term results of tricuspid valve repair and replacement surgery in patients with CIEDs Indeed, patients with TR and CIEDs can be divided in 2 categories: CIEDs induced TR and CIEDs associated TR. In patients with CIEDs induced TR, the valve dysfunction is directly caused by the lead with several mechanism such as mechanical interference with tricuspid valve (TV) leaflet mobility and coaptation (impingement), valve damage during lead placement or manipulation and sub-valvular entanglement. In patients with CIEDs associated TR the valve dysfunction is not directly caused by the lead.

In 2009 approximately 720 000 CIEDs were implanted worldwide [7] and since then a continuous increase of CIEDs implantation was registered, with an estimation of 1.4 millions of CIEDs implantation in 2023. With this impressive number of CIEDs requirement, the need for surgical or trans-catheter treatment of severe TR CIEDs induced or associated, increased steadily in the past years and it likely will continue to increase in the next years. However, limited data are available regarding the outcome of tricuspid valve surgery in patients with CIEDs, particularly for the long-term results. With this study we aim to report the long-term result of tricuspid valve repair and replacement in patients with CIEDs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients;
* Patients with significant, surgically treatable tricuspid regurgitation (TR) according to guidelines
* Patients with an implantable electronic heart device (CIEDs)
* Patients undergoing surgery, both repair or replacement, of the tricuspid valve, both isolated or associated with intervention on the valves of the left heart sections.
* Patients operated at the Cardiac Surgery Department of the San Raffaele Hospital from 2000 to 2019.

Exclusion Criteria:

* Patients without a CIED

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients CIEDs bearer and affected by a surgically treatable tricuspid regurgitation
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2022-02-27 (Actual); Study Completion 2022-02-27 (Actual)

PRIMARY OUTCOMES:
TR recurrency | Through study completion, an average of 7 years

SECONDARY OUTCOMES:
All causes mortality | Through study completion, an average of 7 years
cardiac mortality | Through study completion, an average of 7 years

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No